CLINICAL TRIAL: NCT03891966
Title: Upper Extremity Post-op Splints: Do They Improve Post-operative Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01505
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Extremity Injury
Keywords: Upper Extremity Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint (Active Comparator)
  Interventions: Procedure: Rigid Splint
- Soft Dressing (Active Comparator)
  Interventions: Procedure: Soft Dressing

INTERVENTIONS:
Procedure: Rigid Splint — 50 patients undergoing operative fixation of isolated bothbone forearm, radial head, olecranon, distal humerus, or humeral shaft fractures will either receive a splint.
  Arms: Splint
Procedure: Soft Dressing — 50 patients undergoing operative fixation of isolated both bone forearm, radial head, olecranon, distal humerus, or humeral shaft fractures will either receive a soft dressing post-operatively.
  Arms: Soft Dressing

SUMMARY:
The goal of this study is to determine if applying a rigid splint helps to reduce pain following operative fixation of upper extremity fractures. Orthopedic trauma surgeons currently vary in their application of rigid post-operative splints versus soft dressings after certain surgical procedures based on personal preference. In this study, 100 patients undergoing operative fixation of isolated both bone forearm, radial head, olecranon, distal humerus, or humeral shaft fractures will either receive a splint or soft dressing post-operatively. Their pain, medication usage and function will be tracked over the 2- week postoperative period to see if splinting has any impact on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in study and complete consent
* Will undergo operative fixation of an isolated both bone forearm, radial head, olecranon, distal humerus fracture, or humeral shaft fracture.

Exclusion Criteria:

* Pregnant women
* Patients with concomitant TBI or MR
* Polytrauma patients
* Pathologic Fractures
* Patients undergoing treatment for malignancy
* NYU SoM Students, Residents, Faculty
* Prisoners
* IV drug users or patients on chronic narcotics
* Gun shot wound victims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Percent change in Visual Analog Scale (VAS) | 14 Days
  Best state you can imagine is marked 100and the worst state you can imagine is marked 0 on a line
Percent Change in Euro Quality of Life (EQ-5D) | 14 Days
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Leucht, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Philipp.Leucht@nyulangone.org To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Sgaglione MW, Solasz SJ, Leucht P, Egol KA. Is Postoperative Splinting Advantageous After Upper Extremity Fracture Surgery? Results From the Arm Splint Pain Improvement Research Experiment. J Orthop Trauma. 2024 Mar 1;38(3):e92-e97. doi: 10.1097/BOT.0000000000002742. PMID 38117579